CLINICAL TRIAL: NCT03502668
Title: A Randomized, Open-Label, Phase 1-2 Study of ASTX727 Low Dose (ASTX727 LD) Extended Schedule in Subjects With Lower Risk (IPSS Low or Intermediate-1) Myelodysplastic Syndromes (MDS)
Brief Title: Phase 1-2 Study of Low Dose ASTX727 (ASTX727 LD) in Lower Risk MDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASTX727-03
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: low risk myelodysplastic syndromes, MDS, ASTX727
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine; cedazuridine

STUDY DESIGN:
Intervention Model Description: Multicenter, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Stage A (Experimental): 3 cohorts of 6 subjects each in a schedule in 28-day cycles of ASTX727 LD
  Interventions: Drug: ASTX727 LD
- Phase 1 Stage B (Experimental): 3 cohorts of 10 subjects each in 28-day cycles of ASTX727 LD
  Interventions: Drug: ASTX727 LD
- Phase 2 (Experimental): 80 additional subjects randomized in a 1:1 ratio studying two different doses
  Interventions: Drug: ASTX727 LD; Drug: ASTX727 SD

INTERVENTIONS:
Drug: ASTX727 LD — oral decitabine (LD) + cedazuridine (E7727)
  Other Names: oral decitabine (LD) + cedazuridine (E7727)
Drug: ASTX727 SD — oral decitabine (SD) + cedazuridine (E7727)
  Other Names: oral decitabine (SD) + cedazuridine (E7727)
  Arms: Phase 2

SUMMARY:
Multicenter, open-label study of various ASTX727 LD doses and schedules to assess safety, pharmacodynamics, pharmacokinetics, and hematologic response in subjects with International Prognostic Scoring System (IPSS) risk category of low-risk or Intermediate-1 MDS. This study will be conducted in two phases. In phase 1 subjects will be randomized into 3 cohorts in a 28-day cycles. Phase 2, 80 new subjects will be randomized in a 1:1 ratio into 2 doses/schedules.

DETAILED DESCRIPTION:
A Phase 1-2, multicenter, open-label study of various ASTX727 LD doses and schedules to assess the safety, pharmacodynamics (PD), pharmacokinetics (PK), and hematologic response in subjects with IPSS risk category of low-risk or Intermediate-1 MDS. The study will be conducted in 2 phases.

Phase 1: In Stage A, subjects will be randomized into 3 cohorts of 6 subjects each testing different doses of oral decitabine with cedazuridine in 28-day cycles. When safety has been established in Phase 1 Stage A, Phase 1 Stage B will open, wherein additional 30 subjects will be randomized in a 1:1:1 ratio into 3 cohorts of 10 subjects.

Phase 2: Using 2 doses/schedules one of which will be selected from Phase 1, 40 additional subjects per dose/schedule will be randomized in a 1:1 ratio. The selected doses/schedules will be evaluated for safety (drug-related AEs), efficacy (including hematologic response), PD (long interspersed nucleotide element-1 (LINE-1 methylation, and fetal hemoglobin as fraction of total hemoglobin), and PK.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent before the first study-specific procedure.
2. Men or women ≥18 years with IPSS low risk or Int-1 MDS (all subjects). Subjects must have had at least 1 of the following disease-related criteria during the 8 weeks before randomization:

   1. Red blood cell (RBC) transfusion dependence of 2 or more units of RBC transfusions (RBC transfusion administered for hemoglobin (Hb) levels ≤9.0 g/dL are counted).
   2. Hb of <9.0 g/dL in at least 2 blood counts prior to randomization or in 1 blood count if RBC transfusion was received.
   3. Absolute Neutrophil Count (ANC) of <0.5 × 10^9/L in at least 2 blood counts prior to randomization.
   4. Platelet counts of <50 × 10^9/L in at least 2 blood counts prior to randomization.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
4. Adequate organ function.
5. Women of child-bearing potential (according to recommendations of the Clinical Trial Facilitation Group [CTFG]) must not be pregnant or breastfeeding and must have a negative pregnancy test at screening.
6. Women of child-bearing potential must agree to use contraceptive measures of birth control for 6 months after completing treatment; men must use contraceptive measures and agree not to father a child for at least 3 months after completing treatment.

Exclusion Criteria:

1. Treatment with any investigational drug or therapy within 2 weeks before study treatment.
2. Treatments for MDS must be concluded 1 month prior to study treatment.
3. Prior treatment with azacitidine, decitabine, or guadecitabine.
4. Diagnosis of chronic myelomonocytic leukemia (CMML).
5. Poor medical risk because of other conditions such as uncontrolled systemic diseases or active uncontrolled infections.
6. Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, prostate cancer or breast cancer under control with hormone therapy, or other cancer from which the subject has been disease free for at least 1 year.
7. Known active infection with human immunodeficiency virus or hepatitis viruses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Incidence of drug-related Grade ≥3 Adverse Events (AEs) or dose-limiting toxicities (DLTs) (if any) for each cohort dose/schedule | 18-24 months
  Phase 1: Safety
Hematologic response based on normalization of conversion of any baseline cytopenia or anemia (hemoglobin response, neutrophil response, platelet response, transfusion independence) | 18-24 months
  Phase 2: Efficacy

SECONDARY OUTCOMES:
%LINE-1 methylation change from baseline | 18-24 months
  pharmacodynamics
Area under the curve (AUC) | 18-24 months
  pharmacokinetics parameter
Maximum plasma concentration (Cmax) | 18-24 months
  pharmacokinetics parameter
Time to reach maximum concentration (Tmax) | 18-24 months
  pharmacokinetics parameter
Half life (t1/2) | 18-24 months
  pharmacokinetics parameter
Hematologic response (Phase 1 only) based on normalization of conversion of any baseline cytopenia or anemia (hemoglobin response, neutrophil response, platelet response, transfusion independence) | 18-24 months
  Phase 1: Efficacy
Time to bone marrow blasts >5% | 18-24 months
  Number of days from the date of randomization to the date when bone marrow blasts are >5% and increased by ≥50%.
Leukemia-free survival | 18-24 months
  Number of days from the date of randomization to the date when bone marrow or peripheral blood blasts reach ≥20%, or death from any cause
Overall survival | 18-24 months
  Number of days from the date of randomization to the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (29):
- United States (18):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - University of Colorado, Anschutz Cancer Pavilion, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - BRCR Medical Center Inc., Plantation, Florida
  - Moffitt Cancer Center Site#507, Tampa, Florida
  - The University of Chicago, Chicago, Illinois
  - Indiana University Health Hospital - Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Clinical Research Center, Westwood, Kansas
  - The Center for Cancer and Blood Disorders (RCCA MD LLC - Maryland Division), Bethesda, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Oregon Health and Science University Knight Cancer Institute, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center - Hematology-Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Tyler, Tyler, Texas
- Belgium (2):
  - ZNA - Campus Middelheim, Antwerp
  - Az St-Jan Brugge-Oostende A.V., Bruges
- Canada (2):
  - London Regional Cancer Center, London, Ontario
  - University of Alberta Hospital - Hematology Research, Edmonton
- Germany (2):
  - Universitaetsklinikum Freiburg Site#703, Freiburg im Breisgau
  - Universitätsklinikum Halle, Halle
- Universita degli Studi di Firenze, Florence, Italy
- Spain (4):
  - Hospital Universitario Vall d Hebron, Barcelona
  - Institut Català d'Oncologia Badalona Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Univeristario y Politecnico La Fe Servicio de Hematologia, Valencia

IPD SHARING:
Plan to Share IPD: No